CLINICAL TRIAL: NCT00145912
Title: Primary Care Based Depression Prevention for Adolescents/Young Adults/Young Adults and Young Adults
Acronym: CATCH-IT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: National Alliance for Research on Schizophrenia and Depression (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: C.A.T.C.H.-I.T. - 13240B; 13240B
Record Dates: First submitted 2005-09-01; First posted 2005-09-05 (Estimated); Last update posted 2013-09-05 (Estimated); Status verified 2013-09

CONDITIONS: Depression
Keywords: Depression in adolescents and young adults, depression web-base activity
MeSH Terms: conditions — Depression | interventions — Crisis Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intrinsic Motivation (Experimental): PCP motivational interview + Internet program
  Interventions: Behavioral: MI + CATCH-IT Internet Site
- Extrinsic Motivation (Active Comparator): PCP breif advice + Internet Program
  Interventions: Behavioral: BA (brief advice) + CATCH-IT Internet site

INTERVENTIONS:
Behavioral: MI + CATCH-IT Internet Site — MI + CATCH-IT Internet Site
  Arms: Intrinsic Motivation
Behavioral: BA (brief advice) + CATCH-IT Internet site — BA (brief advice) + CATCH-IT Internet site
  Arms: Extrinsic Motivation

SUMMARY:
The purpose of this research is to evaluate the feasibility of an interview between an adolescent / young adult and a PCP (Primary Care Physician).

DETAILED DESCRIPTION:
A web-based depression prevention program will evaluate the interview. Depression is a condition where people feel sad, tired, have changes in sleep, and lose interest in fun things for more than two weeks. This program teaches adolescents/young adults new skills. They learn new skills by talking with their doctor and doing a workbook at an Internet site. Counselors have used some of these lessons to successfully treat, and in some cases, prevent depression. We do not know if these lessons given in a primary care doctor's office or over the Internet will prevent depression. We will have to do further studies to determine this. If subjects are clinically depressed right now, they cannot be a part of this study.

ELIGIBILITY:
Inclusion Criteria:

* age 15-21 years and
* two risk factors for developing depression in the next two years:

  * Center for Epidemiologic Studies-Depression (CES-D) score > 12 and either a family history or past personal history of depression.
  * Exclusion criteria include meeting criteria or undergoing active treatment for M. depression, or having suicidal ideation

Exclusion Criteria:

* undergoing active treatment for M. depression, or having suicidal ideation

Ages: 15 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 49 (Actual)
Dates: Start 2007-02; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
use of Internet site | 2 months

SECONDARY OUTCOMES:
depressed mood and risk factors | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin W Van Voorhees, MD, Principal Investigator — The University of Chicago, 5841 South Maryland Ave., MC 2007 Chicago, IL 60637
Locations (1):
- The University of Chicago, Chicago, Illinois, United States

REFERENCES:
- [Derived] Eisen JC, Marko-Holguin M, Fogel J, Cardenas A, Bahn M, Bradford N, Fagan B, Wiedmann P, Van Voorhees BW. Pilot Study of Implementation of an Internet-Based Depression Prevention Intervention (CATCH-IT) for Adolescents in 12 US Primary Care Practices: Clinical and Management/Organizational Behavioral Perspectives. Prim Care Companion CNS Disord. 2013;15(6):PCC.10m01065. doi: 10.4088/PCC.10m01065. Epub 2013 Dec 19. PMID 24800110
- [Derived] Hoek W, Marko M, Fogel J, Schuurmans J, Gladstone T, Bradford N, Domanico R, Fagan B, Bell C, Reinecke MA, Van Voorhees BW. Randomized controlled trial of primary care physician motivational interviewing versus brief advice to engage adolescents with an Internet-based depression prevention intervention: 6-month outcomes and predictors of improvement. Transl Res. 2011 Dec;158(6):315-25. doi: 10.1016/j.trsl.2011.07.006. Epub 2011 Aug 19. PMID 22061038
- [Derived] Iloabachie C, Wells C, Goodwin B, Baldwin M, Vanderplough-Booth K, Gladstone T, Murray M, Fogel J, Van Voorhees BW. Adolescent and parent experiences with a primary care/Internet-based depression prevention intervention (CATCH-IT). Gen Hosp Psychiatry. 2011 Nov-Dec;33(6):543-55. doi: 10.1016/j.genhosppsych.2011.08.004. Epub 2011 Sep 28. PMID 21958447